CLINICAL TRIAL: NCT03042819
Title: A Phase 1b Trial of Selinexor Plus Doxorubicin in Advanced Soft Tissue Sarcomas (STS)
Brief Title: Study of Selinexor and Doxorubicin in Advanced Soft Tissue Sarcomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAR-002
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — selinexor; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Selinexor plus Doxorubicin (Experimental): Selinexor will be given by mouth (orally) once a week:
  Dose Level -1 = 40 mg Dose Level 1 (Starting Dose) = 60 mg Dose Level 2 = 80 mg
  Doxorubicin will be given by vein (intravenously) at a dose of 75 mg/m2 once every 3 weeks.
  Interventions: Drug: Selinexor; Drug: Doxorubicin

INTERVENTIONS:
Drug: Selinexor — Selinexor is a Selective Inhibitor of Nuclear Export (SINE) compound that binds and inactivates Exportin 1 (XPO1), thereby forcing the nuclear retention of key tumor suppressor proteins (TSPs).
Drug: Doxorubicin — Doxorubicin is currently approved for various cancers. Doxorubicin inhibits DNA synthesis and repair by inhibiting topoisomerase II and also by intercalation between base pairs on the DNA helix. These actions result in the blockade of DNA and RNA synthesis and fragmentation of DNA.

SUMMARY:
This is a phase 1b study of investigational drug selinexor in combination with doxorubicin in patients with locally advanced or metastatic soft tissue sarcoma. The purpose of this study is to determine how safe and tolerable the combination is, as well as the best dose of the study drugs in this patient population.

Selinexor (also called KPT-330), works by trapping "tumor suppressor proteins" within the cell and thus causing the cancer cells to die or stop growing.

DETAILED DESCRIPTION:
This is a phase 1b study of investigational drug selinexor in combination with doxorubicin in patients with locally advanced or metastatic soft tissue sarcoma.

Patients will be screened for eligibility within 28 days of the start of the study drugs. In addition to standard tests and procedures, research tumor tissue (archival or fresh biopsy) will be collected for collection for pharmacodynamics. Participants will also be asked if they agree to optional biopsies at 6 cycles if their cancer is responding and at disease progression.

Eligible participants will then receive the study drugs in 21 day cycles. Selinexor will be given by mouth and doxorubicin will be given by vein, once a week, for 6 cycles.

Participants will be restaged every 2 cycles. If participants respond to treatment after 6 cycles, they may be able to continue the selinexor alone as a maintenance treatment until progression or unacceptable toxicity.

While receiving the study drug, many of the screening tests will be repeated. Additional tests and procedures include blood sample collection for pharmacokinetics and pharmacodynamics.

When participants stop the study drug permanently for any reason, an end of treatment visit, 28-day follow-up, and long term follow up every 90 days will occur.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* Age ≥ 18 years.
* Patients must have histologically confirmed locally advanced/unresectable or metastatic soft tissue sarcoma.
* Patients must have not received prior doxorubicin.
* Patient must show evidence of progressive disease on study entry or newly diagnosed patients with de novo metastatic measurable disease
* Patient must have measureable disease as defined by RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hematopoietic function
* Adequate hepatic function:
* Adequate renal function
* Adequate cardiac function13
* Patients must agree to use methods of contraception as a agreed upon by the patient and study doctor

Exclusion Criteria:

* Patient is pregnant or lactating
* Radiation, chemotherapy, immunotherapy, any other systemic anticancer therapy, or participation in an investigational anti-cancer study ≤3 weeks prior to initiation of therapy.
* Major surgery within 4 weeks before initiation of therapy
* Unstable cardiovascular function
* Active, ongoing or uncontrolled active infection within one week prior to first dose.
* Malignancies other than disease under study within 2 years prior to Cycle 1, Day 1.
* Known to be HIV seropositive
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or hepatitis B virus (HBV) surface antigen (HBsAg)
* Patients with active CNS malignancy.
* Patients with any gastrointestinal dysfunctions that could interfere with the absorption of Selinexor or patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea.
* Inability or unwillingness to take supportive medications such as anti-nausea and anti anorexia agents.
* In the opinion of the Investigator, patients who are significantly below their ideal body weight
* Serious psychiatric or medical conditions that could interfere with treatment
* Concurrent therapy with approved or investigational anticancer therapeutic agents
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the Incidence of Treatment-Emergent Adverse Events, graded and categorized according to the CTCAE v4.0. | 3 years
  All adverse events will be tabulated and summarized by major organ category, grade, anticipation, and drug attribution. SAE specific incidence and exact 95% confidence interval will be provided where appropriate.
To determine the recommended phase II dose (RP2D) of Selinexor in combination with doxorubicin | 3 years
  The RP2D will be determined according to interim mTPI monitoring algorithm (Figure 5.1) using the dose determining set.

SECONDARY OUTCOMES:
Rate of Grade 3 Toxicities | 3 years
Response Rate | 3 years
Progression-free Survival Rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No